CLINICAL TRIAL: NCT04864626
Title: Study of the Impact on the Evolution of the Disease in the Medium Term of the Implementation of a System of Extended Follow-up by Telephone Interview of Patients With an Eating Disorder Organized by the Nurses of the Eating Disorder Referral Center
Acronym: SPETCA
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 19PH227; 2020-A02830-39 (Other: ANSM)
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-06

CONDITIONS: Eating Disorders; Recurrence; Relapse
MeSH Terms: conditions — Feeding and Eating Disorders; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with eating disorder
  Interventions: Other: semi-standardized interview; Other: care experience questionary

INTERVENTIONS:
Other: semi-standardized interview — annual collection of the number of consultations and hospitalizations at the center, as well as the number of treatments
Other: care experience questionary — questionary with 12 questions to rate the quality of the telephone reception and your feelings during the interview

SUMMARY:
The referral center for eating disorders provides for a systematic many years follow-up of patients under care with an annual assessment at the center. The investigators have recently shown the frequency of relapse in the first 7 years after diagnosis, but the literature remains poor on this epidemiology and on the risk factors for relapse. The investigators would therefore like to extend this follow-up for an additional 3 years after remission with an annual telephone nursing interview for all cured patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with an eating disorder confirmed at the multidisciplinary consultation meeting of the referring center and considered cured (in remission). For patients with Oral Disorders, inclusion is within one year of recovery
* Patient affiliated or entitled to a social security plan
* Oral participation agreement
* Pregnant women

Exclusion Criteria:

* Persons deprived of liberty
* Patients under guardianship or curatorship
* refusal to participate

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient with eating disorders
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of relapses/recurrences per year | 3 years

SECONDARY OUTCOMES:
risk factors for relapse/recurrence | 3 years
  To determinate if one or more factors below could be a risk factors for relapse/recurrence :
  * Age
  * Sex
  * Body mass index
  * Contraception use
  * History of an eating disorder
  * Intense physical activity
  * History of psychiatric hospitalization
  * History of suicide attempt
  * Presence of psychotropic treatment of any kind
Number of patients called per year | 3 years
Number of calls made per patient per year | 3 years
Number of completed calls per patient per year | 3 years
Number of telephone sessions per year per patient | 3 years
Duration of telephone sessions | 3 years
Number of lost to follow-up per year | 3 years
Number of patients not cured | 3 years
Analysis of the experience of care questionnaire | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Marion POY, nurse, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No